CLINICAL TRIAL: NCT01278836
Title: Study of Fasciocutaneous Flaps for Treatment of Leg Defects
Brief Title: Fasciocutaneous Flaps for Leg Defects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Dr. Alireza Yousefy, Associate Professor of Medical Education, Isfahan University of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: ASD-1213-12
Record Dates: First submitted 2011-01-18; First posted 2011-01-19 (Estimated); Last update posted 2011-01-27 (Estimated); Status verified 2009-06

CONDITIONS: Limb Defects
Keywords: Flap; leg defect; reconstruction; tissue

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- fascio-cutaneous flap (Other): flaps which include skin, subcutaneous tissue, and the underlying fascia.
  Interventions: Procedure: fasciocutaneous flap

INTERVENTIONS:
Procedure: fasciocutaneous flap — flaps which include skin, subcutaneous tissue, and the underlying fascia.

SUMMARY:
The purpose of this study is to determine the effects of fasciocutaneous flaps for leg defects.

DETAILED DESCRIPTION:
The fasciocutaneous flaps are tissue flaps which include skin, subcutaneous tissue, and the underlying fascia. Including the deep fascia with its prefascial and subfascial plexus enhances the circulation of these flaps. The investigators determined long-term outcomes of fasciocutaneous flap reconstruction in patients with lower limb defects.

ELIGIBILITY:
Inclusion Criteria:

* patients with leg defects

Exclusion Criteria:

* patients with underlying diseases

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2009-06; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
necrosis | at three years after surgery

SECONDARY OUTCOMES:
venous congestion | at three years after surgery

CONTACTS AND LOCATIONS:
Overall Officials: hamidreza shemshaki, MD, Study Chair — MD,research comittee
Locations (1):
- Kashani University Hospital, Isfahan, Isfahan, Iran